CLINICAL TRIAL: NCT05817240
Title: A Phase 1, Single-Center, Fixed Sequence, Drug-Drug Interaction Study of ENV-101 (Taladegib) on Nintedanib Pharmacokinetics in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study of ENV-101 (Taladegib) on Nintedanib Pharmacokinetics in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endeavor Biomedicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENV-IPF-102
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: smoothened; hedgehog; pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — LY2940680; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: taladegib; Drug: nintedanib

INTERVENTIONS:
Drug: taladegib — 100 mg per tablet, dosed once daily
  Other Names: ENV-101
Drug: nintedanib — 100 mg per capsule, dosed once daily

SUMMARY:
The goal of this clinical trial is to learn about the potential effect of ENV-101 (taladegib) on the pharmacokinetics of nintedanib (an approved treatment for idiopathic pulmonary fibrosis) when the two compounds are dosed together in healthy subjects. Participants in this study will receive ENV-101 and/or nintedanib on various days throughout a 10-day period during which they will reside at the clinical trial site.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥18 and ≤32 kg/m^2
* Body weight ≤120kg
* Subjects must be willing to be sequestered for 10 consecutive days.

Exclusion Criteria:

* Chronic or current use of any prescription medications or acute use within the preceding 30 days or 5 half-lives, whichever is longer, with the exception of contraceptives, prior to study start
* Subject has an active infection of hepatitis B or C, or human immunodeficiency virus (HIV) at study start
* Subject has a history of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers, within 5 years before study start
* Participation in a clinical research trial that included the receipt of an investigational agent or any experimental procedure within 30 days or 5 half-lives, whichever is longer, prior to the screening visit, or planned participation in any such trial at time of study start
* Subject has a pulse <45 or >100 bpm; systolic blood pressure >160 mmHg, or diastolic blood pressure >95 mmHg at study start
* Subject has pacemaker; is not in sinus rhythm; has a corrected QT interval (QTc; using Fridericia's [QTcF] formula) of >450 ms (for males) and >470 ms (for females) during the Screening Period; or has a left bundle branch block or bifascicular block.
* Females and males of reproductive potential who are sexually active and unwilling to use birth control for the duration of the study and for 90 days after their final study dose
* Females that are pregnant or lactating
* Females and males that are unwilling to refrain from blood or blood product donation for the duration of the study and for 30 days after their final study dose
* Males who are unwilling to refrain from sperm donation for the duration of the study and for 90 days after their final study dose
* Females who are unwilling to refrain from egg donation for the duration of the study and for 90 days after their final study dose
* Subjects with a history of a severe allergic reaction or anaphylactic reaction or known hypersensitivity to any component of ENV-101 (taladegib) or nintedanib
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study investigative site or the study Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Nintedanib maximum blood concentration (Cmax) after administration alone and after coadministration with ENV-101 (taladegib) | Day 1 and Day 7
Time of nintedanib maximum blood concentration (Tmax) after coadministration alone and after coadministration with ENV-101 (taladegib) | Day 1 and Day 7
Nintedanib absorption to time t (AUC0-t) after administration alone and after coadministration with ENV-101 (taladegib) | Day 1 and Day 7
  AUC represents "area under the concentration-time curve" and measures the amount of drug that is present in the blood from the time of administration to a given time t
Nintedanib total absorption (AUC0-inf) after administration alone and after coadministration with ENV-101 (taladegib) | Day 1 and Day 7
Nintedanib half-life in the blood (T1/2) after administration alone and after coadministration with ENV-101 (taladegib) | Day 1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Paul Frohna, M.D., Ph.D., Study Director — Endeavor Biomedicines
Locations (1):
- Research Site, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No